CLINICAL TRIAL: NCT00255138
Title: Efficacy of Atomoxetine Therapy Versus Placebo For Ameliorating Cognitive Late Effects Among Survivors of Childhood Cancers
Brief Title: Efficacy of Atomoxetine Therapy Versus Placebo for Cognitive Late Effects
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 4463
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Cancer; Cognitive Late Effects
Keywords: Cancer; Cognitive Late Effects; Stimulants; Atomoxetine; Attention; Children
MeSH Terms: conditions — Neoplasms | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Atomoxetine

SUMMARY:
The purpose of the study is to evaluate the effectiveness and safety of atomoxetine in enhancing attention and concentration among childhood survivors of cancer.

DETAILED DESCRIPTION:
In previous years, it had often been assumed that cognitive and behavioral declines in children who survived cancer therapy were largely a function of the prophylactic therapies (e.g., radiation, chemotherapy) that these children had received. Regardless of the etiologies of these specific late effects, the data regarding the long-term outcome of these children are strikingly consistent. Generally, the studies to date suggest significant impairments in attention and concentration that result in marked declines in academic performance and social and behavior difficulties.

Despite the clear evidence of problems with attention and concentration, as well as associated fucntional impairments (e.g., poor academic achievement and poor peer relationships), there have been few clinical trials designed to manage the cogntive late effects and neurological toxicities associated with radiation therapy and chemotherapy for children and adolescents who have survived cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-18
* Patient has received chemotherapy, radiation, or a combination of both.
* Patient is at least 12 months post-competion of therapy but no more than five years post-completion of therapy.

Exclusion Criteria:

* No ongoing pharmacological management of ADHD
* Not currently pregnant

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2005-11 (Estimated)

PRIMARY OUTCOMES:
Conner's Parent Rating Scale (CPRS)

SECONDARY OUTCOMES:
Conner's Teacher Rating Scale (CTRS)
Continuous Performance Test (CPT)
Side Effects Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ronald T Brown, Ph.D., Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States